CLINICAL TRIAL: NCT06784440
Title: Search for Noninvasive Markers of "Graft Injury" in Pediatric and Adult Patients With Congenital Heart Disease Undergoing Cardiac Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PED-TRANSPLANT-DNA; RC2022 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-12-30; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Congenital Heart Disease (CHD); Heart Transplant Patients; Adult Congenital Heart Disease; Pediatric Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endomyocardial biopsy and analysis for the presence of dd-cfDNA (Other): Whenever a patient enrolled in the study undergoes endomyocardial biopsy, either as part of surveillance of acute myocardial rejection or for clinical suspicion of rejection, concomitantly a blood sample will be taken and analyzed for the presence of dd-cfDNA. In patients with biopsy evidence of acute rejection, a new dd-cfDNA sampling will be performed approximately three months after treatment at the next clinical follow-up
  Interventions: Genetic: Evaluation of circulating donor free DNA in the recipient's blood (Dd-cfDNA: donor-derived cell free DNA)

INTERVENTIONS:
Genetic: Evaluation of circulating donor free DNA in the recipient's blood (Dd-cfDNA: donor-derived cell free DNA) — From the blood samples taken, 2 mL of plasma separated from blood will be stored in EDTA frozen at -80°C. This material will later be processed by NGS run using of CareDX kits. The result will be provided by dedicated software as percentage of donor DNA in relation to recipient DNA.

SUMMARY:
This clinical tissue-based, drug-free, single-center, longitudinal study aims to validate a new diagnostic method, namely, to evaluate whether plasma levels of circulating donor free DNA in the recipient's blood (Dd-cfDNA: donor-derived cell free DNA), in patients undergoing orthotopic heart transplantation, can be predictive of the presence of acute myocardial rejection with the same sensitivity as immunohistochemical analysis on endomyocardial biopsy specimen, the current gold standard for the diagnosis of acute cell-mediated myocardial rejection, in a population consisting of pediatric patients and adult patients with congenital heart disease undergoing orthotopic heart transplantation.

DETAILED DESCRIPTION:
To achieve the study objective, approximately 20 patients of all ages, both pediatric and adult with congenital heart disease and undergoing orthotopic heart transplantation, followed at our center will be enrolled. Whenever a patient enrolled in the study undergoes endomyocardial biopsy, either as part of surveillance of acute myocardial rejection or for clinical suspicion of rejection, concomitantly a blood sample will be taken and analyzed for the presence of dd-cfDNA. In patients with biopsy evidence of acute rejection, a new dd-cfDNA sampling will be performed approximately three months after treatment at the next clinical follow-up. The data collected for each patient will be both baseline anthropometric data and imaging and laboratory variables collected in the normal follow-up provided by clinical practice, as well as data related to the endomyocardial biopsy result and those related to blood sampling for donor DNA.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with congenital heart disease undergoing cardiac transplantation at our center or other centers, followed in follow-up at our center (Unit of Pediatric Cardiology and Developmental Age, IRCCS Azienda Ospedaliero-Universitaria di Bologna)
* Pediatric patients undergoing cardiac transplantation at our center or other centers but followed in follow-up at our center
* Obtaining informed consent from the adult patient or parent/guardian in case of minor

Exclusion Criteria:

* Failure to obtain informed consent from the adult patient or parent/guardian in case of minor

Max Age: 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-11-08 (Estimated); Study Completion 2026-03-07 (Estimated)

PRIMARY OUTCOMES:
Determination of plasma levels of circulating dd-cfDNA in the recipient's blood | 1 day
  The primary aim of this study is to determine whether plasma levels of circulating dd-cfDNA in the recipient's blood can be predictive of the presence of acute myocardial rejection with the same sensitivity as the gold standard represented by immunohistochemical analysis on biopsy specimen. The presence of acute myocardial rejection is defined in accordance with the 2004 ISHLT guidelines as a finding at endomyocardial biopsy of cellulomediated rejection (grade 2R or 3R) and/or humoral rejection (pAMR grade 1,2 or 3), while dd-cfDNA levels, expressed as a percentage relative to the recipient's DNA, will be assessed as pathological both based on the indications in the literature for other forms of rejection (>1%), and as a continuous scale to determine a possible specific cutoff value for our population.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Ragni, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No